CLINICAL TRIAL: NCT03321760
Title: Phase II Evaluation With Safety Run-in of Stereotactic Ablative Body Radiation for T1-2a N1 Non-Small Cell Lung Cancer
Brief Title: SABR for T1-2a N1 NSCLC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Decided not to open the study.
Sponsor: Indiana University (Other)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Principal Investigator, Tim Lautenschlaeger, Assistant Professor of Radiation Oncology, Indiana University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IUSCC-0626; 1707319235 (Other: Indiana University IRB)
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a Phase II single-institution trial with a 3 + 3 safety run-in period. SABR will be delivered per protocol, followed by a planned 4 cycles of sequential chemotherapy within 3-8 weeks after the completion of SABR. Four cycles of chemotherapy shall be planned as typically used for adjuvant chemotherapy following surgical resection for T1-2aN1 non-small cell lung carcinoma (NSCLC) unless otherwise indicated by institutional guidelines.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Run-In Dose 1 (Experimental): 10 Gy dose delivered to the primary tumor & 10 Gy to the hilar (N1) node over 5 fractions
  Interventions: Radiation: Stereotactic Ablative Radiation Therapy (SABR)
- Run-In Dose -1 (Experimental): 10 Gy dose delivered to the primary tumor & 9 Gy to the hilar (N1) node over 5 fractions
  Interventions: Radiation: Stereotactic Ablative Radiation Therapy (SABR)
- Run-In Dose -2 (Experimental): 10 Gy dose delivered to the primary tumor & 8 Gy to the hilar (N1) node over 5 fractions
  Interventions: Radiation: Stereotactic Ablative Radiation Therapy (SABR)
- Phase 2 (Experimental): The maximum tolerated radiation dose to the hilar (N1) node from the run-in period will be used during Phase 2.
  Interventions: Radiation: Stereotactic Ablative Radiation Therapy (SABR)

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiation Therapy (SABR) — SABR will be delivered to the primary disease and hilar (N1) node over 5 fractions.Reductions may be made to the hilar (N1) node according to a 3+3 design during the run-in period.

SUMMARY:
Conventionally fractionated radiation therapy given over 6-7 weeks alone, sequentially, or concurrent with chemotherapy have produced poor outcomes in Stage II NSCLC in most series. Stereotactic ablative radiotherapy (SABR) has been shown to be very effective and is now standard of care for Stage 1 disease. There has been initially reluctance to utilize SABR for central lung tumors because of published reports that showed an excess of toxicity when SABR was utilized; however, newer data with less intense treatment regimens suggest safety in treatment of central lung disease. The safety and efficacy of SABR in treating hilar nodes or N1 disease currently is not known fully and will be evaluated in this study.

DETAILED DESCRIPTION:
1. Primary Objectives Safety run-in - To determine the safety of SABR for the treatment of primary lung disease and N1 (hilar) node in stage T1-2a N1 NSCLC Phase II - To determine 2-year local control of SABR for T1-2a N1 NSCLC with sequential chemotherapy
2. Secondary Objectives Phase II - To determine overall and progression-free survival times, pattern of failures, and rates of ≥ grade 3 adverse events after SABR for T1-2a N1 NSCLC combined with sequential chemotherapy

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years old at time of consent
2. Ability to provide written informed consent and HIPAA authorization
3. Pathological diagnosis of NSCLC lung cancer
4. Staging PET/CT within 45 days of consult
5. EBUS or other histologic confirmation of N1 involvement (diagnosis of lung cancer should come from the hilar [N1] disease)
6. T1/2a <5cm lung primary
7. N1 disease <5cm
8. Patient refuses surgery or deemed inoperable
9. KPS of > 60
10. Baseline labs including CBC/differential and BMP within 45 days of consult
11. CBC/differential with adequate bone marrow function defined as follows:

    1. Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
    2. Platelets ≥ 100,000 cells/mm3
    3. Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.)
12. Adequate renal function defined as serum creatinine within normal institutional limits or creatinine clearance must be at least 20 ml/min
13. Adequate hepatic function defined as total bilirubin ≤ 3.0 x upper limit of normal (ULN) for the institution and ALT, AST, and alkaline phosphatase ≤ 3.0 x ULN for the institution
14. If a pleural effusion is present, the following criteria must be met at registration to exclude malignant involvement (incurable M1a disease):

    1. When pleural fluid is visible on both the CT scan and on a chest x-ray, a pleuracentesis is required to confirm that the pleural fluid is cytologically negative;
    2. Effusions that are minimal (i.e. not visible under ultrasound guidance) and that are too small to safely tap are eligible.
15. Women of childbearing potential and male participants must practice adequate contraception throughout the study
16. Patients with post-obstructive pneumonia are eligible provided they no longer require intravenous antibiotics at registration
17. Eligible for adjuvant chemotherapy as determined by the treating medical oncologist

Exclusion Criteria

1. Previous radiation therapy overlapping with current radiation target as determined by the discretion of the investigator
2. Inability to comply with treatment per investigator discretion.
3. Inability to follow standard of care follow up recommendations per investigator discretion.
4. Pregnant and breastfeeding women
5. Contra-indication to platinum-based two drug chemotherapy as determined by the treating medical oncologist
6. Patients with a history of chronic kidney disease or lactic acidosis
7. Severe, active co-morbidity, defined as follows:

   i. Uncontrolled neuropathy ≥ grade 2 regardless of cause ii. Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months iii. Transmural myocardial infarction within the last 6 months iv. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration v. Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration vi. Severe hepatic disease, defined as a diagnosis of Child-Pugh Class B or C hepatic disease vii. HIV positive with CD4 count < 200 cells/microliter. Note that patients who are HIV positive are eligible, provided they are under treatment with highly active antiretroviral therapy (HAART) and have a CD4 count ≥ 200 cells/microliter within 30 days prior to registration. Note also that HIV testing is not required for eligibility for this protocol.

   viii. End-stage renal disease (i.e. on dialysis or dialysis has been recommended).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of dose-limiting toxicities (DLTs) during the run-in period | 30 days
  Any event per CTCAE v.4 that occurs within 30 days from the start of SABR, and is possibly, probably or definitely related to treatment, and is related to a specific list of symptoms which are outlined in the protocol.

SECONDARY OUTCOMES:
Local control | 2 years
  Failure of disease progression within or immediately adjacent to the treatment planning target volume (PTV) of the lung primary and nodal disease. Failures will be classified as local failures if failing within or immediately adjacent to the N1 or primary tumor PTV, unless judged by the investigator team to convincingly be a separate lesion from the treated lesion (i.e. new lesion within PTV but across a fissure)
Progression free survival | 2 years
  Length of time during and after the treatment that a patient lives with the disease but it does not get worse
Overall survival | 5 years
  Length of time start of treatment that patients are still alive
Rate of dose-limiting toxicities (DLTs) at one year | 1 year
  Any event per CTCAE v.4 that occurs within 1 year from the start of SABR, and is possibly, probably or definitely related to treatment, and is related to a specific list of symptoms which are outlined in the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Lautenschlaeger, MD, Principal Investigator — Indiana University
Locations (3):
- United States (3):
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No